CLINICAL TRIAL: NCT00850161
Title: Intranasal Insulin and Its Effect on Postprandial Glucose Metabolism in Comparison to Subcutaneous Insulin
Brief Title: Intranasal Insulin and Its Effect on Postprandial Metabolism in Comparison to Subcutaneous Insulin
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business purposes.
Sponsor: CPEX Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Nasulin™-BNT-US-100-PK009
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; Nasal Insulin; Insulin Deficiency; Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasulin™ (Experimental): Intranasal insulin spray
  Interventions: Drug: Nasulin™
- aspart (Active Comparator): Subcutaneous administration
  Interventions: Drug: aspart

INTERVENTIONS:
Drug: aspart — Meal-time insulin. Administered subcutaneously based on routine clinical therapy.
  Other Names: insulin aspart
  Arms: aspart
Drug: Nasulin™ — 100 IU(2 puffs in each nostril)
  Other Names: insulin
  Arms: Nasulin™

SUMMARY:
The purpose of this study is to determine if glucose peaks higher and earlier after a meal when a patient is given intranasal insulin instead of conventional insulin treatment.

DETAILED DESCRIPTION:
Diabetes mellitus is a common metabolic disorder characterized by hyperglycemia which when untreated is associated with microvascular disease. Most people with type 1 diabetes are treated with a combination of long-acting (basal) insulin and short-acting (prandial) insulin administered prior to meals. This necessitates multiple daily injections (>3) which is a significant barrier to long-term compliance and treatment. Intranasal administration of insulin has been developed in an effort to overcome the need for insulin injection prior to meals. The pharmacokinetic properties conferred to insulin by this route of administration suggest that postprandial glucose disposal may be stimulated leading to lower glucose concentrations in comparison to dosing via other routes. We propose to study postprandial glucose turnover in healthy volunteers with Type 1 diabetes to determine the effect of intranasal insulin on glucose disposal. We wish to do so in order to develop a greater understanding of how the different bioavailability timing of intranasal insulin might alter postprandial glucose disposal and suppression of endogenous glucose production. In order to address these questions we will address specific aims:

* Peak postprandial glucose disposal is higher and occurs earlier, in the presence of intranasal insulin administration than it is in more conventional forms of insulin dosing.
* Peak suppression of endogenous glucose production is greater and occurs earlier, in the presence of intranasal insulin administration than it is in more conventional forms of insulin dosing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 Diabetes
* Age 18-50
* Treatment management of MDI(multiple daily injections) or Insulin Pump
* BMI between 19-30 Kg/M2
* HbA1c less than or equal to 8.0%
* 75 g OGTT (oral glucose tolerance test)study with insulin concentrations >80uU/mL

Exclusion Criteria:

* Active Proliferative Retinopathy
* Active Nephropathy
* Chronic Upper Respiratory Conditions determined by MD
* Pregnant or Lactating Female

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to determine whether intranasal administration of Nasulin™ will stimulate glucose disposal and suppress endogenous glucose production. | Blood will be measured at -30, -20, -10, 0, 2, 6, 8, 10, 20, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 270, 300, 330 and 360 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No
There is no data; study never initiated.